CLINICAL TRIAL: NCT05103202
Title: Efficacy and Safety of 10-Week or Shorter vs 12-Week or Longer Injection Intervals of Botulinum Toxin for the Treatment of Muscle Spasm Associated With Neurological Disorders
Brief Title: Efficacy and Safety of 10-Week or Shorter vs 12-Week or Longer Injection Intervals of Botulinum Toxin
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Richard Dewey, Professor of Neurology, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0224
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Cervical Dystonia; Blepharospasm; Limb Dystonia; Hemifacial Spasm; Spasticity, Muscle; Fragments of Torsion Dystonia
MeSH Terms: conditions — Torticollis; Blepharospasm; Dystonia; Hemifacial Spasm; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 10 weeks or less: Patients receiving botulinum toxin injections at a frequency of 10 weeks or less
- 12 weeks or more: Patients receiving botulinum toxin injections at a frequency of 12 weeks or more

SUMMARY:
Our hypothesis is that botulinum toxin injections (with onabotulinum toxin, incobotulinum toxin, and abobotulinum toxin) given at 10-week or shorter intervals for the indication of treatment of muscle spasms associated with neurological disorders are associated with equal safety and effectiveness as those given at 12-week or longer intervals. We also hypothesize that for those patients who would prefer a shorter inter-injection interval, but for whom their insurance carrier has prevented this, have worse health-related quality of life compared to patients who receive injections at a 10-week or shorter interval. We aim to investigate this hypothesis by collecting demographic and injection data and patient survey responses.

DETAILED DESCRIPTION:
Our project has the following aims:

Aim 1: to determine if any difference exists in safety or efficacy between patients receiving injections of botulinum toxin at 10-week or shorter intervals as compared to patients receiving injections at 12-week or longer intervals.

Aim 2: to determine if patients who have expressed a preference for injections at 10 week or shorter intervals but whose insurance carriers have mandated a 12-week interval have worse health related quality of life as compared to patients who are receiving injections at 10-week or shorter intervals.

This project consists of two analyses, each designed to accomplish aims 1 and 2. For both aims, we will invite consecutive patients who meet entry criteria to participate who are followed in the botulinum toxin injection clinics of the University of Texas Southwestern Medical Center movement disorders faculty. Participants who consent to data collection by participating in an email-administered survey of quality of life will have their medical records reviewed by an investigator for abstraction of clinical data (to include dose, injection site, injection interval, side effects, demographics, and diagnoses). Additionally, patients will fill out two or more survey instruments on the date of their enrollment visit following their botulinum toxin injection visit. The survey instruments completed will be 1) the SF-36 health questionnaire and 2) a disease-specific HRQoL survey chosen to be applicable to the specific condition for which that subject is receiving botulinum toxin injections. Patients receiving injections for multiple conditions will receive surveys for each condition for which they are receiving treatment. The disease specific scales to be used selectively depending on the patient's specific condition include:

* Blepharospasm disability index
* Craniocervical dystonia questionnaire (CDQ-24)
* Arm dystonia disability scale (ADDS)
* Hemifacial spasm scale (HSF-7)
* Oromandibular dystonia questionnaire (OMDQ-25)
* Spasticity scale (SQoL-6D)

For analysis, patients will be segregated into two groups (10-week or shorter inter-injection interval and 12 week or longer inter-injection interval) on the basis of time elapsed between the most recent botulinum toxin treatments. Clinical and survey data will be analyzed to determine if differences exist between the two groups.

ELIGIBILITY:
Inclusion Criteria

Aim 1:

1. Patient provides responses to an internet based survey which includes consent to participate
2. Patient has been diagnosed with one or more of the conditions for which a HRQoL scale exists and will be employed in this study
3. Patient has received at least 2 prior injections with botulinum toxin for that condition by one of the study investigators
4. Both of the two most recent intervals between injections are either a) 10-weeks or less or b) 12-weeks or more

Aim 2:

1. Patient provides responses to an internet based survey which includes consent to participate
2. Patient has been diagnosed with one or more of the conditions for which a HRQoL scale exists and will be employed in this study
3. Patient has received at least 2 prior injections with botulinum toxin for that condition by one of the study investigators
4. Both of the two most recent intervals between injections are either a) 10-weeks or less or b) 12-weeks or more
5. If receiving injections at 12-weeks or more, notes must have previously indicated that patient needs an injection interval of 10-weeks or less
6. If receiving injections at 12-weeks or more, the reason must be that the insurance carrier covering that patient's medical costs refused to allow a 10-week or less injection frequency

Exclusion Criteria:

For both Aims 1 and 2:

1. Patient is unwilling to consent to study procedures (refuses to fill out surveys)
2. Patient has variable injection frequencies such that the two most recent injections do not both meet criteria of being 10-weeks or less in frequency or 12-weeks or more in frequency
3. Patient has a diagnosis of and is being treated for a condition for which a HRQoL scale does not exist
4. Patient has insufficient chart documentation to characterize demographics, diagnosis, toxin selected, dose used, and injection frequency employed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited consecutively on presentation for treatment of muscle spasm due to neurological disease with botulinum toxin to the UT Southwestern Movement Disorders clinic by one of the investigators.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Quality of Life measured by Short Form 36 (SF-36) | single measure at 1 day of enrollment
  SF-36 HRQoL score as collected by a patient-completed survey (measured from 0 to 100 with a scoring system where 100 is best quality of life)
Safety of injection | single measure at 1 day of enrollment
  Side effects recorded qualitatively and graded by severity (0 to 4 numerical subjective grade where 4 is most severe) by the injecting physician and attributed by that physician to the most recent injection

SECONDARY OUTCOMES:
Blepharospasm disability index survey (BSDI) | single measure at 1 day of enrollment
  Patient-completed survey BSDI- Disease specific quality of life score measured from 0 to 4 calculated as a mean of applicable items with 4 representing worst quality of life
Cervicocranial dystonia questionnaire (CDQ24) | single measure at 1 day of enrollment
  Patient-completed survey CDQ24- Disease specific quality of life score measured from 0 to 100 with 100 representing worst quality of life
Arm Dystonia Disability Scale (ADDS) | single measure at 1 day of enrollment
  Patient-completed survey ADDS- Disease specific quality of life score measured from 0 to 100% with 0% representing worst quality of life
Hemifacial Spasm Scale (HFS7) | single measure at 1 day of enrollment
  Patient-completed survey HFS7- Disease specific quality of life score (measured from 0 to 4 where 4 is the most severe effect on quality of life)
Oromandibular dystonia questionnaire (OMDQ-25) | single measure at 1 day of enrollment
  Patient-completed survey OMDQ-25- Disease specific quality of life score (measured from 0 to 100 with 100 representing worst quality of life)
Spasticity Quality of Life scale (SQoL-6D) | single measure at 1 day of enrollment
  Patient-completed survey SQoL-6D- Disease specific quality of life score (measured from 0 to 100 with 100 representing best quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dewey, Jr., MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson DM, Hallett M, Ashman EJ, Comella CL, Green MW, Gronseth GS, Armstrong MJ, Gloss D, Potrebic S, Jankovic J, Karp BP, Naumann M, So YT, Yablon SA. Practice guideline update summary: Botulinum neurotoxin for the treatment of blepharospasm, cervical dystonia, adult spasticity, and headache [RETIRED]: Report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2016 May 10;86(19):1818-26. doi: 10.1212/WNL.0000000000002560. Epub 2016 Apr 18. PMID 27164716
- [Background] Tan EK, Fook-Chong S, Lum SY, Thumboo J. Validation of a short disease specific quality of life scale for hemifacial spasm: correlation with SF-36. J Neurol Neurosurg Psychiatry. 2005 Dec;76(12):1707-10. doi: 10.1136/jnnp.2005.065656. PMID 16291898
- [Background] Wissel J. Towards flexible and tailored botulinum neurotoxin dosing regimens for focal dystonia and spasticity - Insights from recent studies. Toxicon. 2018 Jun 1;147:100-106. doi: 10.1016/j.toxicon.2018.01.018. Epub 2018 Jan 31. PMID 29407165
- [Background] Truong DD, Gollomp SM, Jankovic J, LeWitt PA, Marx M, Hanschmann A, Fernandez HH; Xeomin US Blepharospasm Study Group. Sustained efficacy and safety of repeated incobotulinumtoxinA (Xeomin((R))) injections in blepharospasm. J Neural Transm (Vienna). 2013 Sep;120(9):1345-53. doi: 10.1007/s00702-013-0998-9. Epub 2013 Feb 23. PMID 23435927
- [Background] Evidente VG, Truong D, Jankovic J, Comella CL, Grafe S, Hanschmann A. IncobotulinumtoxinA (Xeomin(R)) injected for blepharospasm or cervical dystonia according to patient needs is well tolerated. J Neurol Sci. 2014 Nov 15;346(1-2):116-20. doi: 10.1016/j.jns.2014.08.004. Epub 2014 Aug 10. PMID 25186131
- [Background] Greene P, Fahn S, Diamond B. Development of resistance to botulinum toxin type A in patients with torticollis. Mov Disord. 1994 Mar;9(2):213-7. doi: 10.1002/mds.870090216. PMID 8196686
- [Background] Jankovic J, Vuong KD, Ahsan J. Comparison of efficacy and immunogenicity of original versus current botulinum toxin in cervical dystonia. Neurology. 2003 Apr 8;60(7):1186-8. doi: 10.1212/01.wnl.0000055087.96356.bb. PMID 12682332
- [Background] Ruta D, Garratt A, Abdalla M, Buckingham K, Russell I. The SF 36 health survey questionnaire. A valid measure of health status.. BMJ. 1993 Aug 14;307(6901):448-9. doi: 10.1136/bmj.307.6901.448-b. No abstract available. PMID 8374477
- [Background] Jankovic J, Kenney C, Grafe S, Goertelmeyer R, Comes G. Relationship between various clinical outcome assessments in patients with blepharospasm. Mov Disord. 2009 Feb 15;24(3):407-13. doi: 10.1002/mds.22368. PMID 19053054
- [Background] Muller J, Wissel J, Kemmler G, Voller B, Bodner T, Schneider A, Wenning GK, Poewe W. Craniocervical dystonia questionnaire (CDQ-24): development and validation of a disease-specific quality of life instrument. J Neurol Neurosurg Psychiatry. 2004 May;75(5):749-53. doi: 10.1136/jnnp.2003.013441. PMID 15090572
- [Background] Peterson DA, Berque P, Jabusch HC, Altenmuller E, Frucht SJ. Rating scales for musician's dystonia: the state of the art. Neurology. 2013 Aug 6;81(6):589-98. doi: 10.1212/WNL.0b013e31829e6f72. Epub 2013 Jul 24. PMID 23884039
- [Background] Fahn, S., Assessment of the primary dystonias, in Quantification of Neurologic Deficit, M. TL, Editor. 1989, Butterworths: Oxford. p. 241-270.
- [Background] Merz RI, Deakin J, Hawthorne MR. Oromandibular dystonia questionnaire (OMDQ-25): a valid and reliable instrument for measuring health-related quality of life. Clin Otolaryngol. 2010 Oct;35(5):390-6. doi: 10.1111/j.1749-4486.2010.02194.x. PMID 21108749
- [Background] Turner-Stokes L, Ashford S, Jacinto J, Maisonobe P, Balcaitiene J, Fheodoroff K. Impact of integrated upper limb spasticity management including botulinum toxin A on patient-centred goal attainment: rationale and protocol for an international prospective, longitudinal cohort study (ULIS-III). BMJ Open. 2016 Jun 17;6(6):e011157. doi: 10.1136/bmjopen-2016-011157. PMID 27315835